CLINICAL TRIAL: NCT03710148
Title: The Effect of Iodine Intakes on Maternal and Infant Health and the Study of Iodine RNI for Different Stages of Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wanqi Zhang (Other)
Collaborators: Shandong Institute for Endemic Disease Control and Research (Unknown); Tianjin Maternal and Child Health Care Center (Unknown)
Responsible Party: Sponsor-Investigator, Wanqi Zhang, Vice Dean for School of Public Health, Tianjin Medical University
Organization: Tianjin Medical University (Other)
Other Study IDs: NSFC-81330064
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Iodine Reaction; Iodine Compounds Overdose; Pregnancy Related
Keywords: Iodine; Estimated Average Requirement; Recommended Nutritent Intake; Tolerable Upper Intake Level; Pregnant Women; Pregnancy; EAR; RNI; UL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Natural exposure of deficient or excessive iodine — Natural exposure of deficient iodine from diet & drinking water, and of excessive iodine intake from drinking water

SUMMARY:
This study determined the effects of different iodine intake on the maternal and infant health and provide evidence for studying the RNI and UL of iodine in pregnant women.

1. The study of effect on mothers and their infants of the lack of iodine at different gestation in adequate iodine area.

   The purpose of this study was to detect the maternal thyroid function, growth and neuropsychological development of infants in different pregnancy women with diverse iodine intake levels, and to make a clear evaluation for the influence of iodine deficiency during different pregnancy by following up iodine suitable early pregnancy women and mild iodine deficient three pregnancy women as well as their infants.
2. The study of recommended iodine intake (RNI) for healthy pregnant women in three pregnancy.

   Different pregnancy women with different iodine intake levels were recruited and carried out iodine balance experiment in the case of not interfering with their diet. In addition, the iodine intake of the pregnant women when they reached "zero iodine balance" was calculated, that was EAR of iodine in pregnant women. In conclusion, the iodine balance experiment in pregnant women at different pregnancy improved the sample collection methods and evaluation criteria and was more scientific and reasonable than the classic iodine balance experiment.
3. The study of effect of different levels of high iodine exposure on pregnant women, delivery women and their infants.

In this study, we made a prospective study of the early pregnancy women and their infants exposed to different high iodine levels in high water iodine areas. At first we defined the effects of long-term iodine excess exposure on the health of the mother and the infants by combining with the reference index of the normal value of the thyroid function in different maternal and postpartum periods, the level of growth and development of the offspring and the assessment of the level of neuropsychological development. Furthermore the harmful effects of different high levels of iodine exposure on pregnant women was synthetically analyzed. This study obtained the safe intake level of iodine for pregnant women and provided scientific basis for the formulation of iodine UL in pregnant women in China.

DETAILED DESCRIPTION:
1. The relationship between iodine deficiency during pregnancy and maternal offspring health

1. Screening of pregnant women with iodine deficiency:

   A prevalence survey of pregnant women was conducted in iodine-sufficient area, combined with the results of single spot urinary concentration, 24h urinary iodine concentration and thyroglobulin level, screening out pregnant women with iodine deficiency during first, second and third trimester of pregnancy. There are 60 pregnant women in each group. At the same time, 60 pregnant women with iodine-sufficient during early pregnancy were selected, and the total number of the four groups is 240.
2. Effects of iodine deficiency on pregnant women during different pregnancy:

   Pregnant women with iodine deficiency were gived nutritional guidance, and were advised to take iodine supplements. Follow-up with regularly collecting fasting venous blood, dried whole blood and single spot urine was conducted, in order to dynamically grasp the iodine nutritional status and thyroid function of pregnant women during different pregnancy, and clarify the influence of iodine deficiency on pregnant women in each group.
3. Effects of iodine deficiency on offspring during different pregnancy:

   The offspring of follow-up pregnant women were observed, collecting the heel blood at birth for measuring TSH, and performing physical examination. Assessment of neuropsychological development in offspring for two years after delivery was performed , in order to clarify the effects of iodine deficiency on the neuropsychological development of offspring in each group.
4. Statistical analysis:

Normally distributed variables were reported as the mean ± standard deviation, comparison between groups were analyzed with the use of t-test or analysis of variance (ANOVA), and Pearson linear correlation was used for correlation analysis; Urinary iodine level is lognormal distribution, so it was converted into logarithmic form and then analyzed. Non-normally distributed variables were presented as median and interquartile range. The Wilcoxon rank sum test was used for comparison between groups, and correlation analysis was performed using the Spearman rank correlation test. The chi-squared test was adopted for the comparison of enumeration data. P values below 0.05 was considered statistically significant.

2. Study the RNI of iodine on pregnant women during different pregnancy:

1. Screening of pregnant women during different pregnancy:

   A prevalence survey of pregnant women was conducted in iodine-sufficient area, based on 24h urinary iodine concentration, thyroglobulin level, related health check and medical history query results, screening out pregnant women who meet the requirements of this study during first, second and third trimester of pregnancy. Each group has 20 pregnant women, and the total number is 60.
2. Reasearch of the iodine EAR of pregnant women during different pregnancy:

   Iodine balance studies were performed on healthy pregnant women during first, second and third trimester of pregnancy to evaluate the daily iodine intake and excretion, including collecting and testing 24h dietary iodine intake, 24h urinary iodine and fecal iodine excretion of subjects. The daily respiratory iodine intake and excretion of subjects was assessed by measuring the iodine content in the air and exhaled breath. In addition, according to the positive correlation between iodine balance value and iodine intake, a scatter plot was drawn and curve fitting was performed. According to the results of iodine balance experiment, the iodine balance regression curves of first, second and third trimester of pregnancy were established , in order to determine the level of iodine intake when the pregnant women reach the iodine balance, which is the estimated average requirement (EAR) of pregnant women during different pregnancy.
3. Research of iodine RNI on pregnant women during different pregnancy:

Based on the obtained EAR values of iodine for different pregnancy and the 20% coefficient of variation (CV), according to the formula: RNI=EAR+2CV=1.4EAR, the iodine RNI values of pregnant women in different gestation were derived.

3. Study on the relationship between iodine excess and maternal offspring health and iodine UL of pregnant women

1. Prospective study:

   Pregnant women during early pregnancy who were exposed to different excessive water iodine intake were enrolled in a large-scale epidemiological prospective study, in order to assess the levels of iodine intake by collecting and testing random urinary iodine and 24h urinary iodine levels, and to detect the thyroid function indicators under different iodine intake levels to evaluate the health effects and harms of different high iodine intake on pregnant women. At the same time, the growth and development of the offspring and the level of neuropsychological development were evaluated to determine the long-term iodine excess exposure to the health of pregnant women and offspring.
2. Discussion on iodine UL of pregnant women:

   According to the urinary iodine level during pregnancy, the subjects were divided into groups with different iodine intakes, with the TSH abnormal rate of pregnant women > 5% and the increase of FT3/FT4 as the end point, comprehensively determining the harmful effects of different iodine intake on pregnant women and offspring, analyzing the iodine safety intake level suitabled for pregnant women, and exploring the iodine UL of pregnant women.
3. Statistical methods:

Epi-data was used to enter survey data. Univariate statistical analysis was used to analyze the differences in evaluation indicators between different iodine intake levels.. Multivariate statistical analysis methods were used to analyze the safety of each iodine intake level under multiple factors.

ELIGIBILITY:
Inclusion Criteria:

* 1) aged between 18-35 years old; 2) singleton pregnancy; 3) Living in Tianjin or Shandong at least 5 years; 4) no history of any thyroid diseases; 5) no medication or supplementation of iodine.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women were recruited at Tanggu Maternity Hospital and Maternal, Tianjin Child Health Care Service Center and the Maternal and Gaoqing Child Health Hospital, Shandong.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Thyroid goiter confirmed by ultrasonographic thyroid volume | 3 years
  Thyroid lobe volume was calculated according to the following formula: V (mL)=0.479×d×w×l (mm)/1000, and TV was records as the sum of both lobes.
Thyroid dysfunction confirmed by serum concentrations of FT3, FT4, TSH ,TPOAB and TGAb | 3 years
  Thyroid function is not in the normal reference range and is defined as thyroid dysfunction
Evaluation of neuropsychological development of children at age 2 | 2 years
  Children were tested by the neurodevelopmental scale compiled by the Capital Institute of Pediatrics.In this experiment, DQ (> 130) was classified as excellent, 115-129 as upper, 85-114 as middle, 70-84 as lower, and (< 69) as mental retardation.
Iodine intake were measured by Iodine balance experiment | 1 years
  24h iodine intake =24h dietary iodine intake + 24h water iodine intake + 24h respiratory iodine intake

CONTACTS AND LOCATIONS:
Overall Officials: Ping Shao, Master, Principal Investigator — Tianjin Maternal and Child Health Care Center; Xiaoming Wang, Master, Principal Investigator — Shandong Institute for Endemic Disease Control and Research; Laixing Lin, Master, Principal Investigator — Tianjin Medical University Metabolic Diseases Hospital; Jun Shen, Master, Principal Investigator — Tianjin Medical University; Long Tan, PhD, Principal Investigator — Tianjin Medical University; Wen Chen, PhD, Principal Investigator — Tianjin Medical University; Wei Wang, BA, Principal Investigator — Tianjin Medical University; Tingkai Cui, BA, Principal Investigator — Tianjin Medical University; Min Gao, BA, Principal Investigator — Tianjin Medical University; Yanting Chen, BA, Principal Investigator — Tianjin Medical University; Wenxing Guo, BA, Principal Investigator — Tianjin Medical University; Chongdan Wang, BA, Principal Investigator — Tanggu Maternity Hospital
Locations (3):
- China (3):
  - Gaoqing Maternal and Child Health Care Center, Zibo, Shandong
  - Tanggu Maternity Hospital, Tianjin
  - Tianjin Maternal and Child Health Care Center, Tianjin

REFERENCES:
- [Background] Sang Z, Wang PP, Yao Z, Shen J, Halfyard B, Tan L, Zhao N, Wu Y, Gao S, Tan J, Liu J, Chen Z, Zhang W. Exploration of the safe upper level of iodine intake in euthyroid Chinese adults: a randomized double-blind trial. Am J Clin Nutr. 2012 Feb;95(2):367-73. doi: 10.3945/ajcn.111.028001. Epub 2011 Dec 28. PMID 22205314
- [Background] Boyages SC. Clinical review 49: Iodine deficiency disorders. J Clin Endocrinol Metab. 1993 Sep;77(3):587-91. doi: 10.1210/jcem.77.3.8370679. No abstract available.
- [Background] Zimmermann MB, Andersson M. Update on iodine status worldwide. Curr Opin Endocrinol Diabetes Obes. 2012 Oct;19(5):382-7. doi: 10.1097/MED.0b013e328357271a. PMID 22892867
- [Background] Caldwell KL, Makhmudov A, Ely E, Jones RL, Wang RY. Iodine status of the U.S. population, National Health and Nutrition Examination Survey, 2005-2006 and 2007-2008. Thyroid. 2011 Apr;21(4):419-27. doi: 10.1089/thy.2010.0077. PMID 21323596
- [Background] Hollowell JG, Haddow JE. The prevalence of iodine deficiency in women of reproductive age in the United States of America. Public Health Nutr. 2007 Dec;10(12A):1532-9; discussion 1540-1. doi: 10.1017/S1368980007360862. PMID 18053275
- [Background] Fuse Y, Ohashi T, Yamaguchi S, Yamaguchi M, Shishiba Y, Irie M. Iodine status of pregnant and postpartum Japanese women: effect of iodine intake on maternal and neonatal thyroid function in an iodine-sufficient area. J Clin Endocrinol Metab. 2011 Dec;96(12):3846-54. doi: 10.1210/jc.2011-2180. Epub 2011 Sep 28. PMID 21956426
- [Background] Vandevijvere S, Amsalkhir S, Mourri AB, Van Oyen H, Moreno-Reyes R. Iodine deficiency among Belgian pregnant women not fully corrected by iodine-containing multivitamins: a national cross-sectional survey. Br J Nutr. 2013 Jun 28;109(12):2276-84. doi: 10.1017/S0007114512004473. Epub 2012 Oct 19. PMID 23084115
- [Background] Zou S, Wu F, Guo C, Song J, Huang C, Zhu Z, Yu H, Guo Y, Lu X, Ruan Y. Iodine nutrition and the prevalence of thyroid disease after salt iodization: a cross-sectional survey in Shanghai, a coastal area in China. PLoS One. 2012;7(7):e40718. doi: 10.1371/journal.pone.0040718. Epub 2012 Jul 27. PMID 22911705
- [Background] Swanson CA, Zimmermann MB, Skeaff S, Pearce EN, Dwyer JT, Trumbo PR, Zehaluk C, Andrews KW, Carriquiry A, Caldwell KL, Egan SK, Long SE, Bailey RL, Sullivan KM, Holden JM, Betz JM, Phinney KW, Brooks SP, Johnson CL, Haggans CJ. Summary of an NIH workshop to identify research needs to improve the monitoring of iodine status in the United States and to inform the DRI. J Nutr. 2012 Jun;142(6):1175S-85S. doi: 10.3945/jn.111.156448. Epub 2012 May 2. PMID 22551802
- [Background] Zimmermann M, Delange F. Iodine supplementation of pregnant women in Europe: a review and recommendations. Eur J Clin Nutr. 2004 Jul;58(7):979-84. doi: 10.1038/sj.ejcn.1601933. PMID 15220938
- [Background] Brucker-Davis F, Ferrari P, Gal J, Berthier F, Fenichel P, Hieronimus S. Iodine status has no impact on thyroid function in early healthy pregnancy. J Thyroid Res. 2012;2012:168764. doi: 10.1155/2012/168764. Epub 2012 Nov 28. PMID 23251828
- [Background] Zimmermann MB. The adverse effects of mild-to-moderate iodine deficiency during pregnancy and childhood: a review. Thyroid. 2007 Sep;17(9):829-35. doi: 10.1089/thy.2007.0108. PMID 17956157
- [Background] Delange F. Iodine requirements during pregnancy, lactation and the neonatal period and indicators of optimal iodine nutrition. Public Health Nutr. 2007 Dec;10(12A):1571-80; discussion 1581-3. doi: 10.1017/S1368980007360941. PMID 18053281
- [Background] Burns R, O'Herlihy C, Smyth PP. The placenta as a compensatory iodine storage organ. Thyroid. 2011 May;21(5):541-6. doi: 10.1089/thy.2010.0203. Epub 2011 Mar 21. PMID 21417918
- [Background] Lazarus JH. Thyroid function in pregnancy. Br Med Bull. 2011;97:137-48. doi: 10.1093/bmb/ldq039. Epub 2010 Dec 23. PMID 21186204
- [Background] Institute of Medicine (US) Panel on Micronutrients. Dietary Reference Intakes for Vitamin A, Vitamin K, Arsenic, Boron, Chromium, Copper, Iodine, Iron, Manganese, Molybdenum, Nickel, Silicon, Vanadium, and Zinc. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222310/ PMID 25057538
- [Background] Delange F, Burgi H. Iodine deficiency disorders in Europe. Bull World Health Organ. 1989;67(3):317-25. PMID 2670299
- [Background] Yu KW, Chin NX, Neu HC. Comparative in vitro activity and beta-lactamase stability of RU29246, the active metabolite of HR916B. Eur J Clin Microbiol Infect Dis. 1992 Jul;11(7):652-9. doi: 10.1007/BF01961678. PMID 1396779
- [Background] Berghout A, Wiersinga W. Thyroid size and thyroid function during pregnancy: an analysis. Eur J Endocrinol. 1998 May;138(5):536-42. doi: 10.1530/eje.0.1380536. PMID 9625365
- [Background] Romano R, Jannini EA, Pepe M, Grimaldi A, Olivieri M, Spennati P, Cappa F, D'Armiento M. The effects of iodoprophylaxis on thyroid size during pregnancy. Am J Obstet Gynecol. 1991 Feb;164(2):482-5. doi: 10.1016/s0002-9378(11)80004-9. PMID 1992688
- [Background] Glinoer D. Iodine supplementation during pregnancy: importance and biochemical assessment. Exp Clin Endocrinol Diabetes. 1998;106 Suppl 3:S21. doi: 10.1055/s-0029-1212040. No abstract available. PMID 9865548
- [Background] Dworkin HJ, Jacquez JA, Beierwaltes WH. Relationship of iodine ingestion to iodine excretion in pregnancy. J Clin Endocrinol Metab. 1966 Dec;26(12):1329-42. doi: 10.1210/jcem-26-12-1329. No abstract available. PMID 5959526
- [Background] Teng W, Shan Z, Teng X, Guan H, Li Y, Teng D, Jin Y, Yu X, Fan C, Chong W, Yang F, Dai H, Yu Y, Li J, Chen Y, Zhao D, Shi X, Hu F, Mao J, Gu X, Yang R, Tong Y, Wang W, Gao T, Li C. Effect of iodine intake on thyroid diseases in China. N Engl J Med. 2006 Jun 29;354(26):2783-93. doi: 10.1056/NEJMoa054022. PMID 16807415
- [Background] Laurberg P, Bulow Pedersen I, Knudsen N, Ovesen L, Andersen S. Environmental iodine intake affects the type of nonmalignant thyroid disease. Thyroid. 2001 May;11(5):457-69. doi: 10.1089/105072501300176417. PMID 11396704
- [Background] Dunn JT. Iodine should be routinely added to complementary foods. J Nutr. 2003 Sep;133(9):3008S-10S. doi: 10.1093/jn/133.9.3008S. PMID 12949401
- [Background] Moon S, Kim J. Iodine content of human milk and dietary iodine intake of Korean lactating mothers. Int J Food Sci Nutr. 1999 May;50(3):165-71. doi: 10.1080/096374899101201. PMID 10627832
- [Background] Andersson M, Karumbunathan V, Zimmermann MB. Global iodine status in 2011 and trends over the past decade. J Nutr. 2012 Apr;142(4):744-50. doi: 10.3945/jn.111.149393. Epub 2012 Feb 29. PMID 22378324
- [Background] Leung AM, Pearce EN, Braverman LE. Iodine nutrition in pregnancy and lactation. Endocrinol Metab Clin North Am. 2011 Dec;40(4):765-77. doi: 10.1016/j.ecl.2011.08.001. PMID 22108279
- [Background] Mao IF, Ko YC, Chen ML. The stability of iodine in human sweat. Jpn J Physiol. 1990;40(5):693-700. doi: 10.2170/jjphysiol.40.693. PMID 2086989
- [Derived] Wang Y, Tian X, Song Q, Wang W, Guo X, Cui T, Pan Z, Chen Y, Chen W, Tan L, Zhang W. Application and Comparison of Different Regression Models in Iodine Balance Experiment on Women of Childbearing Age and Pregnant Women. Biol Trace Elem Res. 2024 Jun;202(6):2474-2487. doi: 10.1007/s12011-023-03867-x. Epub 2023 Oct 9. PMID 37807000
- [Derived] Wu W, Chen Y, Guo W, Zhang K, Chen W, Fu M, Pan Z, Yang Y, Zhang N, Zhang W. The Relationship Between Iodine Excess and Thyroid Function During Pregnancy and Infantile Neurodevelopment at 18-24 Months. J Nutr. 2023 Aug;153(8):2320-2327. doi: 10.1016/j.tjnut.2023.05.012. Epub 2023 May 12. PMID 37182695
- [Derived] Chen W, Wang W, Gao M, Chen Y, Guo W, Dong S, Sun H, Pan Z, Pearce EN, Tan L, Shen J, Zhang W. Iodine Intakes of <150 mug/day or >550 mug/day are Not Recommended during Pregnancy: A Balance Study. J Nutr. 2023 Jul;153(7):2041-2050. doi: 10.1016/j.tjnut.2022.10.017. Epub 2022 Dec 22. PMID 37100687